CLINICAL TRIAL: NCT00434408
Title: Impact of Umbilical Cord Cleansing With Chlorhexidine on Neonatal Mortality and Omphalitis in Rural Sylhet District of Bangladesh
Brief Title: Impact of Umbilical Cord Cleansing With 4.0% Chlorhexidine on Neonatal Mortality
Acronym: CHX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Government of Bangladesh (Other Government); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Save the Children (Other); Shimantik (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB00000146; GHSA00030001900 (Other Grant/Funding Number: Save the Children 131)
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2022-10-05 (Actual); Status verified 2007-07

CONDITIONS: Omphalitis; Infection
Keywords: omphalitis; neonates; umbilical cord; infection; infant mortality; neonate morbidity; chlorhexidine
MeSH Terms: conditions — Infections; Infant Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 4.0% chlorhexidine cleansing of the cord during home visits by project workers for the first 7 days after birth
  Interventions: Behavioral: CHX x 7 days
- 2 (Experimental): 4.0% chlorhexidine cleansing of the cord applied once by a project worker visiting the newborn in the home as soon as possible after birth
  Interventions: Behavioral: chx once
- 3 (Active Comparator): dry cord care
  Interventions: Behavioral: dry cord care

INTERVENTIONS:
Behavioral: chx once — 4.0% chlorhexidine cleansing of the cord applied once by a project worker visiting the newborn in the home as soon as possible after birth
  Arms: 2
Behavioral: CHX x 7 days — 4.0% chlorhexidine cleansing of the cord during home visits by project workers for the first 7 days after birth
  Arms: 1
Behavioral: dry cord care — Household members are instructed to apply nothing to the newborn's umbilical cord stump.
  Arms: 3

SUMMARY:
A community based trial that seeks to address the effect of umbilical cord cleansing using 4.0% chlorhexidine cleansing solution

DETAILED DESCRIPTION:
Of the annual four million neonatal deaths, 99% occur in developing countries, and more than one-third globally can be attributed to infections. In areas with high-mortality rates, the proportion attributable to infections is as high as 50%. Many infections in infants can be prevented or treated with already existing measures, yet finding the best way to provide these measures in communities that are limited in resources need to be identified. Applying chlorhexidine to the umbilical cord of newborns may be a simple way to help reduce neonatal mortality and morbidity in the community at low cost.

A study by our group was recently completed in Nepal. It was a large community-based, factorial-designed trial in southern Nepal to: (1) assess the impact of newborn total body skin cleansing with 0.25% chlorhexidine on neonatal mortality and morbidity and (2) assess the impact of cleansing of the umbilical stump with 4% chlorhexidine on omphalitis and neonatal mortality.

The results of these studies have suggested that chlorhexidine antisepsis interventions may significantly reduce neonatal mortality and omphalitis. A single full body cleansing of the neonate with chlorhexidine as soon as possible after birth reduced mortality among low birth weight (LBW) infants by 28%. Repeated cleansing of the umbilical stump with chlorhexidine reduced the rate of severe cord infection by 75% and, if this treatment was begun within the first 24 hours following birth, reduced neonatal mortality by 34%.

In rural Bangladesh, over 90% of women deliver at home with only untrained local women or family members in attendance, and low birth weight babies are delivered approximately 30% of the time. The overall neonatal mortality rate exceeds 36 per 1000 live births and in order to reduce this burden, simple, cost-effective interventions that can be delivered at the community level are urgently needed. Given the potential impact of repeated chlorhexidine cleansing of the cord demonstrated in the Nepal trial, a replication study of this regimen and further investigations of more simple regimens are necessary. The number of treatments necessary to reduce neonatal mortality has important programmatic implications for who can deliver the intervention, and how it is packaged.

ELIGIBILITY:
Inclusion Criteria:

* live-born infants delivered in one of three upazillas of Sylhet District (Zakiganj, Khanaighat, Beanibazar)
* married women of reproductive age within their individual target areas listed above

Exclusion Criteria:

* individuals outside of the target area in Sylhet(Zakiganj, Khanaighat, Beanibazar)
* infants not met at home by a project worker during the first seven days of life

Ages: 1 Minute to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28797 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
neonatal mortality | 3 Month intervals
omphalitis among live born infants. | 3 Month intervals

SECONDARY OUTCOMES:
newborn care practices | 3 Years
care seeking behaviors | 3 Years
morbidity measures, including sepsis and omphalitis | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah H Baqui, MBBS, DrPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Shams El Arifeen, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Rural Sylhet District, Sylhet, Bangladesh

REFERENCES:
- [Background] Aggett PJ, Cooper LV, Ellis SH, McAinsh J. Percutaneous absorption of chlorhexidine in neonatal cord care. Arch Dis Child. 1981 Nov;56(11):878-80. doi: 10.1136/adc.56.11.878. PMID 7305432
- [Background] Baqui AH, Darmstadt GL, Williams EK, Kumar V, Kiran TU, Panwar D, Srivastava VK, Ahuja R, Black RE, Santosham M. Rates, timing and causes of neonatal deaths in rural India: implications for neonatal health programmes. Bull World Health Organ. 2006 Sep;84(9):706-13. doi: 10.2471/blt.05.026443. PMID 17128340
- [Background] Darmstadt GL, Bhutta ZA, Cousens S, Adam T, Walker N, de Bernis L; Lancet Neonatal Survival Steering Team. Evidence-based, cost-effective interventions: how many newborn babies can we save? Lancet. 2005 Mar 12-18;365(9463):977-88. doi: 10.1016/S0140-6736(05)71088-6. PMID 15767001
- [Background] Lawn JE, Cousens S, Zupan J; Lancet Neonatal Survival Steering Team. 4 million neonatal deaths: when? Where? Why? Lancet. 2005 Mar 5-11;365(9462):891-900. doi: 10.1016/S0140-6736(05)71048-5. PMID 15752534
- [Background] Mullany LC, Darmstadt GL, Khatry SK, Katz J, LeClerq SC, Shrestha S, Adhikari R, Tielsch JM. Topical applications of chlorhexidine to the umbilical cord for prevention of omphalitis and neonatal mortality in southern Nepal: a community-based, cluster-randomised trial. Lancet. 2006 Mar 18;367(9514):910-8. doi: 10.1016/S0140-6736(06)68381-5. PMID 16546539
- [Background] Mullany LC, Darmstadt GL, Tielsch JM. Safety and impact of chlorhexidine antisepsis interventions for improving neonatal health in developing countries. Pediatr Infect Dis J. 2006 Aug;25(8):665-75. doi: 10.1097/01.inf.0000223489.02791.70. PMID 16874163
- [Derived] Mitra DK, Mullany LC, Harrison M, Mannan I, Shah R, Begum N, Moin MI, El Arifeen S, Baqui AH; Projahnmo Study Group in Bangladesh. Incidence and risk factors of neonatal infections in a rural Bangladeshi population: a community-based prospective study. J Health Popul Nutr. 2018 Mar 9;37(1):6. doi: 10.1186/s41043-018-0136-2. PMID 29523194
- [Derived] Mullany LC, Shah R, El Arifeen S, Mannan I, Winch PJ, Hill A, Darmstadt GL, Baqui AH. Chlorhexidine cleansing of the umbilical cord and separation time: a cluster-randomized trial. Pediatrics. 2013 Apr;131(4):708-15. doi: 10.1542/peds.2012-2951. Epub 2013 Mar 18. PMID 23509175
- [Derived] Arifeen SE, Mullany LC, Shah R, Mannan I, Rahman SM, Talukder MR, Begum N, Al-Kabir A, Darmstadt GL, Santosham M, Black RE, Baqui AH. The effect of cord cleansing with chlorhexidine on neonatal mortality in rural Bangladesh: a community-based, cluster-randomised trial. Lancet. 2012 Mar 17;379(9820):1022-8. doi: 10.1016/S0140-6736(11)61848-5. Epub 2012 Feb 8. PMID 22322124
- [Derived] Mullany LC, El Arifeen S, Winch PJ, Shah R, Mannan I, Rahman SM, Rahman MR, Darmstadt GL, Ahmed S, Santosham M, Black RE, Baqui AH. Impact of 4.0% chlorhexidine cleansing of the umbilical cord on mortality and omphalitis among newborns of Sylhet, Bangladesh: design of a community-based cluster randomized trial. BMC Pediatr. 2009 Oct 21;9:67. doi: 10.1186/1471-2431-9-67. PMID 19845951